CLINICAL TRIAL: NCT07126366
Title: COLOR STABILITY OF S-PRG RESIN-BASED LIGHT CURE VARNISH AND PROPHYLAXIS PASTE ON WHITE SPOT LESIONS: A 12-MONTH RANDOMIZED CLINICAL TRIAL
Brief Title: Color Stability of S-PRG Resin-Based Light-Cure Varnish and Prophylaxis Paste on White Spot Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy hassan aref abdelaziz, Dr. Engy Hassan Aref, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14422023489475
Record Dates: First submitted 2025-06-27; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: White Spot Lesion of Tooth
Keywords: S-PRG; White spot lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-PRG-Barrier coat ,Shofu Inc. Kyoto, Japan (Active Comparator): A light-cured Giomer varnish for prolonged hypersensitivity relief. Seals and protects exposed dentinal tubules to prevent pain. Ideal for patients experiencing loss of enamel, gingival recession or temporary sensitivity due to whitening.
  Interventions: Other: S-PRG Barrier coat
- S-PRG PROPHYLAXIS PASTE (Experimental): S-PRG PROPHYLAXIS PASTE is a bioactive Giomer-based paste containing S-PRG particles that release six therapeutic ions-fluoride, strontium, borate, aluminum, sodium, and silicate each contributing to remineralization, antibacterial effects, and dentin sensitivity reduction.
  Interventions: Other: S-PRG Prophylaxis paste

INTERVENTIONS:
Other: S-PRG Barrier coat — A light-cured Giomer varnish for prolonged hypersensitivity relief. Seals and protects exposed dentinal tubules to prevent pain. Ideal for patients experiencing loss of enamel, gingival recession or temporary sensitivity due to whitening.
  Arms: S-PRG-Barrier coat ,Shofu Inc. Kyoto, Japan
Other: S-PRG Prophylaxis paste — S-PRG Prophylaxis paste is a bioactive Giomer-based paste containing S-PRG particles that release six therapeutic ions-fluoride, strontium, borate, aluminum, sodium, and silicate each contributing to remineralization, antibacterial effects, and dentin sensitivity reduction.
  Arms: S-PRG PROPHYLAXIS PASTE

SUMMARY:
The aim of the study is to evaluate and compare the long-term color stability of two bioactive materials used in the management of white spot lesions: Surface Pre-Reacted Glass (S-PRG) containing resin-based light-cured varnish and S-PRG containing prophylaxis paste. The study will assess color changes over a 12-month period to determine which material better maintains aesthetic integrity while providing therapeutic benefits for demineralized enamel surfaces.

DETAILED DESCRIPTION:
White spot lesions (WSLs), particularly prevalent in post-orthodontic patients (up to 96%), pose both aesthetic and pathological challenges due to subsurface enamel demineralization that alters optical properties. Although fluoride-based remineralization therapies can arrest lesion progression, they often fail to restore the natural appearance of enamel, leaving residual opacity.

Surface Pre-Reacted Glass (S-PRG) technology offers a bioactive alternative, releasing multiple therapeutic ions (e.g., fluoride, strontium, silicate) to enhance remineralization, neutralize acids, and exhibit antibacterial effects. S-PRG materials are available in resin-based varnishes and prophylaxis pastes; however, their long-term color stability remains underexplored.

Given that aesthetic outcomes significantly impact patient satisfaction, this study aims to compare the 12-month color stability of S-PRG resin-based varnish versus S-PRG prophylaxis paste. Color changes may result from water sorption, dietary staining, polymer degradation, and ion interaction with oral fluids. The comparison is clinically relevant as both materials utilize the same bioactive core but differ in formulation and application methods.

A 12-month observation period allows assessment under real oral conditions, including pH fluctuations and staining challenges. Objective color evaluation using CIE Lab* values and spectrophotometry ensures standardized, clinically relevant data. The study targets anterior teeth due to their aesthetic significance and addresses a critical gap in the literature, supporting evidence-based selection of materials that balance therapeutic efficacy with long-term aesthetic outcomes in WSL management.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting in the outpatient clinic.
* Enamel caries in anterior permanent teeth according to ICDAS-1 and ICDAS-2.
* Good oral hygiene.
* Provide informed consent.
* Cooperative and willing to participate in the trial.
* Male or female.
* Adult patients aged 16 to 35 years.

Exclusion Criteria:

* Spontaneous or elicited pain from caries.
* Tooth mobility.
* Signs of pulpal infection.
* Severe medical conditions that would not allow management in the clinic.
* Hereditary developmental defects such as amelogenesis imperfecta or dentinogenesis imperfecta.
* Known allergies or sensitivities to dental materials, including fluoride
* Inability to return for recall visits.
* Poor oral hygiene.
* Refusal to participate in the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Visual assessment using ICDAS criteria at baseline, 3, 6, and 12 months | at baseline, 3 months, 6 months and 12 months
  Primary Outcome Measure 1:
  Title: Visual Caries Assessment Using ICDAS Criteria Description: Visual/tactile examination of white spot lesions according to the International Caries Detection and Assessment System (ICDAS).
  Score 0: No visible caries (sound tooth)
  Score 1: First visual change in enamel (white or brown opacity, visible only when dry)
  Score 2: Distinct visual change in enamel (opacity visible wet and dry)
  Score 3: Localized enamel breakdown (no visible dentin)
  Score 4: Underlying dark shadow from dentin (no cavitation)
  Score 5: Distinct cavity with visible dentin
  Score 6: Extensive cavity with visible dentin Time Frame: Baseline, 3 months, 6 months, 12 months Unit of Measure: ICDAS score (ordinal scale: 0-6)

SECONDARY OUTCOMES:
Color stability measured by spectrophotometric analysis (ΔE values) at baseline, 3, 6, and 12 months. | at baseline, 3 months,6 months and 12 months
  Color stability measured by spectrophotometric analysis (ΔE values) at baseline, 3, 6, and 12 months.
  Clinical success rate (ΔE ≤ 3.7)
Patient satisfaction scores (VAS 0-10) Color stability measured by spectrophotometric analysis (ΔE values) at baseline, 3, 6, and 12 months Clinical success rate (ΔE ≤ 3.7) | at baseline, 3 months,6 months and 12 months
  Patient satisfaction scores (VAS 0-10) Color stability measured by spectrophotometric analysis (ΔE values) at baseline, 3, 6, and 12 months Clinical success rate (ΔE ≤ 3.7) -